CLINICAL TRIAL: NCT05627258
Title: VRC 615: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB-0115-AB (VRC01.23LS), Administered Intravenously or Subcutaneously to Healthy Adults
Brief Title: A Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRCHIVMAB0115-00-AB (VRC01.23LS), Administered Intravenously or Subcutaneously to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10000889; 000889-I
Record Dates: First submitted 2022-11-23; First posted 2022-11-25 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-09-18

CONDITIONS: HIV
Keywords: Monoclonal Antibody; CD4 Binding; HIV envelope; First in Human; Broadly Neutralizing

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 5 mg/kg IV single administration
  Interventions: Biological: VRC-HIVMAB0115-00-AB
- Group 2 (Experimental): 5 mg/kg SC single administration
  Interventions: Biological: VRC-HIVMAB0115-00-AB
- Group 3 (Experimental): 20 mg/kg IV single administration
  Interventions: Biological: VRC-HIVMAB0115-00-AB
- Group 4 (Experimental): 40 mg/kg IV single administration
  Interventions: Biological: VRC-HIVMAB0115-00-AB
- Group 5 (Experimental): 5 mg/kg SC repeat dosing
  Interventions: Biological: VRC-HIVMAB0115-00-AB
- Group 6 (Experimental): 20 mg/kg IV repeat dosing
  Interventions: Biological: VRC-HIVMAB0115-00-AB

INTERVENTIONS:
Biological: VRC-HIVMAB0115-00-AB — VRC01.23LS, a broadly neutralizing monoclonal antibody targeting the HIV-1 envelope CD4 binding site.

SUMMARY:
Background:

HIV causes AIDS, a serious disease that can lead to fatal infections. HIV infection can be controlled but not cured, nor is there a vaccine to prevent it. Antibodies may offer a promising new way to prevent HIV infection. Antibodies are proteins that are naturally made by the body to fight germs. One antibody (VRC01.23LS) has been tested in the lab and was found to block HIV-like viruses. Researchers want to find out if it is safe to inject VRC01.23LS into people.

Objective:

To test the safety of VRC01.23LS in healthy adults.

Eligibility:

Healthy people aged 18 to 60 years.

Design:

Participants were divided into 6 groups:

Some got 1 dose of VRC01.23LS. They visited the clinic up to 14 times in 24 weeks.

Some got 3 doses, each 12 weeks apart. They had 25 clinic visits over 48 weeks.

For some participants, the drug was given through a tube attached to a needle inserted into a vein in the arm. This took about 30 to 90 minutes. Others received the drug as an injection under the skin in a fatty area of the belly, arm, or thigh; each dose may have needed up to 3 individual injections.

Participants stayed in the clinic up to 8 hours on the days they received VRC01.23LS.

Participants received a thermometer and measuring tool. They checked their temperature daily for 7 days after they received the study drug. They measured any redness, swelling, or bruising at the injection site.

DETAILED DESCRIPTION:
Study Design:

This first-in-human, open-label study evaluated VRC01.23LS (VRCHIVMAB0115- 00-AB) in a dose-escalation design to examine safety, tolerability, dose, and pharmacokinetics (PK) in healthy adults. The primary hypothesis was that subcutaneous (SC) and intravenous (IV) administrations of VRC01.23LS will be safe and well-tolerated in healthy adults. A secondary hypothesis was that VRC01.23LS will be detectable in human sera with a definable half-life.

Study Products:

The VRC01.23LS broadly neutralizing monoclonal antibody (bnAb) targets the CD4 binding site in the HIV-1 envelope, is human in origin, and contains two amino acid modifications within the C-terminus of the heavy chain constant region designed to improve the antibody half-life in vivo. VRC01.23LS was developed by the VRC/NIAID/NIH and manufactured under cGMP regulations at the VRC Pilot Plant operated under contract by the Vaccine Clinical Materials Program (VCMP), Leidos Biomedical Research, Inc., Frederick. MD.

Subjects:

Healthy adults, 18-60 years of age

Study Plan:

This open-label study included 6 groups to evaluate VRC01.23LS administered as a single dose or as repeated doses, given 12 weeks apart as shown in the table below. Enrollment began with the 5 mg/kg dose groups, and enrollment in subsequent dose groups proceeded after dose-escalation safety reviews. Assessment of safety included solicited reactogenicity, clinical observation, and monitoring of hematological and metabolic parameters at clinical visits throughout the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

1. Willing and able to complete the informed consent process.
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
3. Available for clinical follow-up through the last study visit.
4. 18 to 60 years of age.
5. In good general health without clinically significant medical history.
6. Physical examination without clinically significant findings within the 56 days prior to enrollment.
7. Adequate venous access if assigned to an IV group or adequate abdominal subcutaneous tissue if assigned to SC group.
8. Willing to have blood samples collected, stored indefinitely, and used for research purposes.

   Laboratory Criteria within 56 days prior to enrollment:
9. White blood cell count (WBC): 2,500-12,000/mm3.
10. WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
11. Platelets: 125,000 - 500,000/mm3.
12. Hemoglobin within institutional normal range or accompanied by PI or designee approval.
13. Creatinine: <= 1.1 x Upper Limit of Normal (ULN).
14. ALT: <= 1.25 x ULN.
15. AST: <= 1.25 x ULN.
16. Negative for HIV infection by an FDA approved method of detection.

    Female-Specific Criteria:
17. Agrees to use an effective means of birth control from 21 days prior to enrollment through the duration of study participation.
18. Negative Beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply:

1. Woman who is breast-feeding or planning to become pregnant during study participation.
2. Weight > 115 kg.
3. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study.
4. Hypertension that is not well controlled.
5. Receipt of any investigational study product within 28 days prior to enrollment (Note: Emergency Use Authorization of a COVID-19 vaccine is not exclusionary).
6. Receipt of an investigational HIV vaccine or anti-HIV monoclonal antibody.
7. Receipt of any live attenuated vaccine within 28 days prior to enrollment.
8. Receipt of any vaccine within 2 weeks prior to enrollment.
9. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
10. Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, infectious disease, autoimmune disease, psychiatric disorder, heart disease, or cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesia K Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Please refer to protocol Section 9.3.4.

REFERENCES:
- [Background] Gaudinski MR, Coates EE, Houser KV, Chen GL, Yamshchikov G, Saunders JG, Holman LA, Gordon I, Plummer S, Hendel CS, Conan-Cibotti M, Lorenzo MG, Sitar S, Carlton K, Laurencot C, Bailer RT, Narpala S, McDermott AB, Namboodiri AM, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 606 Study Team. Safety and pharmacokinetics of the Fc-modified HIV-1 human monoclonal antibody VRC01LS: A Phase 1 open-label clinical trial in healthy adults. PLoS Med. 2018 Jan 24;15(1):e1002493. doi: 10.1371/journal.pmed.1002493. eCollection 2018 Jan. PMID 29364886
- [Background] Gaudinski MR, Houser KV, Doria-Rose NA, Chen GL, Rothwell RSS, Berkowitz N, Costner P, Holman LA, Gordon IJ, Hendel CS, Kaltovich F, Conan-Cibotti M, Gomez Lorenzo M, Carter C, Sitar S, Carlton K, Gall J, Laurencot C, Lin BC, Bailer RT, McDermott AB, Ko SY, Pegu A, Kwon YD, Kwong PD, Namboodiri AM, Pandey JP, Schwartz R, Arnold F, Hu Z, Zhang L, Huang Y, Koup RA, Capparelli EV, Graham BS, Mascola JR, Ledgerwood JE; VRC 605 study team. Safety and pharmacokinetics of broadly neutralising human monoclonal antibody VRC07-523LS in healthy adults: a phase 1 dose-escalation clinical trial. Lancet HIV. 2019 Oct;6(10):e667-e679. doi: 10.1016/S2352-3018(19)30181-X. Epub 2019 Aug 28. PMID 31473167
- [Background] Kwon YD, Asokan M, Gorman J, Zhang B, Liu Q, Louder MK, Lin BC, McKee K, Pegu A, Verardi R, Yang ES, Program VP, Carlton K, Doria-Rose NA, Lusso P, Mascola JR, Kwong PD. A matrix of structure-based designs yields improved VRC01-class antibodies for HIV-1 therapy and prevention. MAbs. 2021 Jan-Dec;13(1):1946918. doi: 10.1080/19420862.2021.1946918. PMID 34328065
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000889-I.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: VRC-HIVMAB0115-00-AB: VRC01.23LS - 5 mg/kg IV single administration
- Group 2: VRC-HIVMAB0115-00-AB: VRC01.23LS - 5 mg/kg SC single administration
- Group 3: VRC-HIVMAB0115-00-AB: VRC01.23LS - 20 mg/kg IV single administration
- Group 4: VRC-HIVMAB0115-00-AB: VRC01.23LS - 40 mg/kg IV single administration
- Group 5: VRC-HIVMAB0115-00-AB: VRC01.23LS - 5 mg/kg SC repeat dosing, 3 times 12 weeks apart
- Group 6: VRC-HIVMAB0115-00-AB: VRC01.23LS - 20 mg/kg IV repeat dosing, 3 times 12 weeks apart
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Started | 4 | 3 | 3 | 3 | 5 | 5
Completed Product Administration (One (1) participant in Group 5 had mild, self-limiting (Grade 1) creatinine elevation after the 2nd dose and the team decided not to administer the 3rd dose. Two (2) participants in Group 6 did not receive the third dose per the Sponsor's decision to terminate product administration due to safety concerns (occurrence of palpitations in several participants).) | 3 | 3 | 3 | 3 | 2 | 3
Completed | 1 | 3 | 2 | 3 | 3 | 5
Not Completed | 3 | 0 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Enrolled, but product not administered | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other subject illness/injury | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subject moved from area | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 3: VRC-HIVMAB0115-00-AB: VRC01.23LS- 20 mg/kg IV single administration
- Group 5: VRC-HIVMAB0115-00-AB: VRC01.23LS - 5 mg/kg SC repeat dosing:3 times, 12 weeks apart
- Group 6: VRC-HIVMAB0115-00-AB: VRC01.23LS - 20 mg/kg IV repeat dosing: 3 times, 12 weeks apart
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 5 | 5 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (3.2) | 44.3 (7.1) | 21.3 (0.6) | 28.7 (12.2) | 26.2 (4.3) | 29.6 (5.6) | 29.3 (8.4)
Age, Customized [Count of Participants; unit: Participants]
  AGE: Ages 18-20 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  AGE: Ages 21-30 | 3 | 0 | 3 | 1 | 4 | 2 | 13
  AGE: Ages 31-40 | 1 | 1 | 0 | 0 | 1 | 3 | 6
  AGE: Ages 41-60 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 2 | 2 | 3 | 11
  Male | 2 | 2 | 2 | 1 | 3 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 3 | 2 | 2 | 2 | 5 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 0 | 1 | 4
  White | 2 | 1 | 1 | 2 | 3 | 4 | 13
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 68.0 (16.8) | 82.9 (11.4) | 66.7 (11.7) | 75.2 (18.3) | 81.7 (26.9) | 68.6 (11.00) | 73.8 (17.1)
Education [Count of Participants; unit: Participants]
  Less than a high school graduate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  High school graduate/GED | 0 | 0 | 0 | 1 | 1 | 0 | 2
  College/University | 4 | 2 | 3 | 1 | 3 | 3 | 16
  Advanced degree | 0 | 1 | 0 | 1 | 1 | 2 | 5
  Not Collected | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Participants recorded the occurrence of solicited local symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017)
Time Frame: 7 days after product administration
Population: Population included all enrolled participants who received study product and provided safety data (via diary card and/or laboratory results) following vaccine administration (N=22). One participant in Group 1 did not receive study product due to onset of a panic attack after IV insertion.
Measure: Count of Participants; unit: Participants
Groups:
- Group 5: VRC-HIVMAB0115-00-AB: VRC01.23LS -5 mg/kg SC repeat dosing: 3 times 12, weeks apart
- Group 6: VRC-HIVMAB0115-00-AB: VRC01.23LS - 20 mg/kg IV repeat dosing: 3 times 12, weeks apart
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
Participants
  Pain/Tenderness: None | 3 | 2 | 2 | 3 | 3 | 4
  Pain/Tenderness: Mild | 0 | 1 | 1 | 0 | 1 | 1
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 1 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 3 | 2 | 2 | 3 | 5 | 5
  Swelling: Mild | 0 | 0 | 1 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 1 | 0 | 0 | 0 | 0
  Redness: None | 3 | 2 | 2 | 3 | 3 | 5
  Redness: Mild | 0 | 0 | 1 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 2 | 0
  Redness: Severe | 0 | 1 | 0 | 0 | 0 | 0
  Pruritus: None | 3 | 2 | 2 | 3 | 3 | 5
  Pruritus: Mild | 0 | 0 | 1 | 0 | 2 | 0
  Pruritus: Moderate | 0 | 1 | 0 | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: None | 3 | 3 | 1 | 3 | 4 | 5
  Bruising: Mild | 0 | 0 | 2 | 0 | 1 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 3 | 1 | 1 | 3 | 1 | 4
  Any Local Symptom: Mild | 0 | 1 | 2 | 0 | 1 | 1
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 3 | 0
  Any Local Symptom: Severe | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Participants recorded the occurrence of solicited systemic symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017
Time Frame: 7 days after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 5: VRC-HIVMAB0115-00-AB: VRC01.23LS - 5 mg/kg SC repeat dosing: 3 times, 12 weeks apart
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
Participants
  Malaise: None | 3 | 3 | 3 | 2 | 2 | 3
  Malaise: Mild | 0 | 0 | 0 | 0 | 3 | 1
  Malaise: Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 2 | 3 | 3 | 3 | 2 | 4
  Myalgia: Mild | 1 | 0 | 0 | 0 | 3 | 1
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 3 | 3 | 3 | 2 | 2 | 3
  Headache: Mild | 0 | 0 | 0 | 1 | 3 | 2
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 3 | 2 | 4 | 3
  Chills: Mild | 0 | 0 | 0 | 0 | 1 | 2
  Chills: Moderate | 0 | 0 | 0 | 1 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 2 | 3 | 3 | 2 | 4 | 3
  Nausea: Mild | 1 | 0 | 0 | 0 | 1 | 2
  Nausea: Moderate | 0 | 0 | 0 | 1 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 3 | 3 | 5 | 5
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 3 | 3 | 3 | 3 | 5 | 5
  Joint Pain: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 2 | 3 | 3 | 1 | 1 | 2
  Any Systemic Symptom: Mild | 1 | 0 | 0 | 1 | 4 | 2
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events Following Product Administration
Description: SAEs were recorded from receipt of product administration through the last study visit at Week 24 for participants in Groups 1, 2, 3, 4. SAEs were recorded from receipt of product administration through the last study visit at Week 48 for participants in Groups 5 or 6. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after product administration through Day 168, up to Week 24 for participants in Groups 1-4. Day 0 after product administration through Day 336, up to Week 48, for participants in Group 5 and 6.
Population: Population included all enrolled participants who received study product (N=22). One participant in Group 1 did not receive study product due to onset of a panic attack after IV insertion.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0 | 0 | 0
  Total Number of Participants who had SAE | 0 | 0 | 0 | 0 | 0 | 0
  Total number of Participants who did not have SAE | 3 | 3 | 3 | 3 | 5 | 5

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Product Administration
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of study product administration through the visit scheduled for 4 weeks after study product administration. At other time periods greater than 4 weeks after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 28 days post product administration, up to Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
participants
  Related to Study Product | 0 | 0 | 1 | 3 | 2 | 2
  Unrelated to Study Product | 0 | 0 | 1 | 0 | 1 | 0
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 0 | 0 | 2 | 3 | 3 | 2
  Total Number of Participants who had no Unsolicited AEs | 3 | 3 | 1 | 0 | 2 | 3

5. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of study product administration through the last expected study visit at Week 24 for Groups 1-4 and through Week 48 for Groups 5-6. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after product administration through Day 140, up to Week 24 for Groups 1-4. Day 0 after product administration through Day 336, up to Week 48 for Groups 5-6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants With New Chronic Medical Condition | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants With No New Chronic Medical Condition | 3 | 3 | 3 | 3 | 5 | 5

6. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following Product Administration
Description: Abnormal lab results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included pregnancy test, hematology and chemistry labs, and HIV Serology diagnostic test. Institutional lab normal ranges as well as the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 - July 2017 were used.
Time Frame: Day 0 after product administration through Day 140, up to Week 24 for Groups 1-4. Day 0 after product administration through Day 336, up to Week 48, for Groups 5-6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
Participants
  Bilirubin | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0 | 1 | 0
  Number of Participants With No Abnormal lab results recorded as unsolicited adverse events (AEs) | 3 | 3 | 3 | 2 | 4 | 5

7. Secondary Outcome: Pharmacokinetic (PK) Parameters of VRC01.23LS: Maximum Observed Serum Concentration (Cmax)
Description: Cmax is the peak serum concentration that VRC01.23LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
Time Frame: Baseline through 24 weeks after VRC01.23LS product administration
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Group 5/ Dose 1; Group 5/ Dose 2; Group 5/ Dose 3: VRC-HIVMAB0115-00-AB: VRC01.23LS - 5 mg/kg SC repeat dosing
- Group 6/Dose 1; Group 6/Dose 2; Group 6/Dose 3: VRC-HIVMAB0115-00-AB: VRC01.23LS - 20 mg/kg IV repeat dosing
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5/ Dose 1 | Group 5/ Dose 2 | Group 5/ Dose 3 | Group 6/Dose 1 | Group 6/Dose 2 | Group 6/Dose 3
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 2 | 5 | 5 | 3
mcg/mL | 96.4 (9.7) | 13.4 (3.9) | 343.5 (51.7) | 719.8 (109.7) | 14.1 (5.4) | 12.9 (5.1) | 19 (5.9) | 428 (60.9) | 491 (61) | 437 (85)

8. Secondary Outcome: Pharmacokinetic (PK) Parameters of VRC01.23LS: Time to Reach Maximum Observed Serum Concentration (Tmax)
Description: Tmax is the time it takes to reach Cmax of VRC01.23LS after it has been administered; it is determined based on the summary PK curve for each dose group.
Time Frame: Baseline through 24 weeks after VRC01.23LS product administration
Measure: Mean (Standard Deviation); unit: days
Groups:
- Group 3: VRC-HIVMAB0115-00-AB: VRC01.23LS -20 mg/kg IV single administration
- Group 5/ Dose 1: VRC-HIVMAB0115-00-AB: VRC01.23LS- 5 mg/kg SC repeat dosing
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5/ Dose 1 | Group 5/ Dose 2 | Group 5/ Dose 3 | Group 6/Dose 1 | Group 6/Dose 2 | Group 6/Dose 3
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 2 | 5 | 5 | 3
days | 0.024 (0.003) | 2.9 (0.011) | 0.024 (0.001) | 0.042 (0.019) | 2.7 (0.42) | 2.9 (0) | 4 (1.4) | 0.023 (0.001) | 0.032 (0.021) | 0.039 (0.013)

9. Secondary Outcome: Pharmacokinetic (PK) Parameters of VRC01.23LS: Beta Half-life (T1/2b)
Description: Beta half-life (T1/2b) is the time required for half of the VRC01.23LS product to be eliminated from the serum.
Time Frame: Baseline through 24 weeks after VRC01.23LS product administration
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5
days | 27.2 (1.8) | 43.3 (9.8) | 51.4 (3.2) | 53.6 (4.3) | 53.3 (26.9) | 40.9 (4)

10. Secondary Outcome: Pharmacokinetic (PK) Parameters of VRC01.23LS: Clearance Rate
Description: Clearance is the rate of VRC01.23LS elimination divided by the plasma VRC01.23LS concentration; determined based on the summary pharmacokinetic (PK) curve for each study group. Clearance following a SC administration is calculated as Clearance (CL)/Bioavailability (F).
Time Frame: Baseline through 24 weeks after VRC01.23LS product administration
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
mL/day | 395.6 (61.6) | 667.5 (43.8) | 478.2 (81.1) | 504.4 (94.1) | 688 (255.9) | 458.1 (88.2)

11. Secondary Outcome: Pharmacokinetic (PK) Parameters of VRC01.23LS: Volume of Distribution
Description: Theoretical volume that would be necessary to contain the total amount of administered drug at the same concentration as observed in plasma. It represents the degree to which a drug is distributed in body tissue rather than the plasma and calculated based in the PK curve for each study group. Volume of distribution following a SC administration is calculated as Volume of distribution (V)/Bioavailability (F).
Time Frame: Baseline through 24 weeks after VRC01.23LS product administration
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5
L | 14.7 (1.6) | 38.2 (6.9) | 32.3 (3.7) | 35.6 (4.2) | 44.7 (40.7) | 24.7 (3.9)

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after product administration. Unsolicited AEs were reported for 4 weeks after study product administration. Serious AEs and new chronic medical conditions were reported through last study visit (up to Week 24 for Groups 1-4 and up to 48 weeks for Groups 5 and 6).
Description: The overall Arms/Groups summarize AEs collected after product administration separately and grouped by the study product and dose. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity. Influenza/ILI were collected separately and not included as AE.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 3/3 | 3/3 | 4/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=3) | Group 2 (N=3) | Group 3 (N=3) | Group 4 (N=3) | Group 5 (N=5) | Group 6 (N=5)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (4)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 2 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 2 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Administration site pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (8) | 1 (1)
Administration site swelling (General disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 0 (0) | 1 (4) | 1 (5) | 0 (0) | 2 (3) | 0 (0)
Administration site prurituis (General disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Administration site bruising (General disorders) | 0 (0) | 0 (0) | 2 (14) | 0 (0) | 1 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT05627258/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT05627258/ICF_000.pdf